CLINICAL TRIAL: NCT03258658
Title: A Phase 1 Pilot Safety and Feasibility Study of Autologous Engineered Urethral
Brief Title: Safety and Feasibility Study of Autologous Engineered Urethral Constructs for the Treatment of Strictures
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00043624; 40010001209 (Other Grant/Funding Number: California Inst. for Regenerative Med)
Record Dates: First submitted 2017-08-03; First posted 2017-08-23 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Urologic Diseases; Male Urogenital Diseases; Urethral Stricture; Urethral Injury
Keywords: Urethral Stricture
MeSH Terms: conditions — Urologic Diseases; Male Urogenital Diseases; Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous Engineered Urethral Construct (Experimental): All subjects enrolled will undergo a full-thickness bladder biopsy as an out-patient surgical procedure. Urothelial and Smooth Muscle Cells recovered from the biopsy will be isolated and expanded over the next 4-6 weeks, and then seeded onto a tubular scaffold to create the autologous engineered urethral construct. Subjects will undergo a second surgical procedure to excise the urethral stricture and implant the urethral construct. All subjects will be followed for 3 years for safety and efficacy.
  Interventions: Biological: Autologous Engineered Urethral Construct

INTERVENTIONS:
Biological: Autologous Engineered Urethral Construct — urethral construct

SUMMARY:
This is a Phase I clinical study to determine the safety and efficacy of using autologous, engineered urethral constructs for the treatment of urethral strictures in adult males.

The proposed study design is a prospective non-randomized and uncontrolled single-center investigation. Autologous urothelial cells (UCs) and smooth muscle cells (SMCs), obtained from enrolled male subjects' bladder tissue samples, will be culture expanded in vitro and used to seed tubular PGA scaffolds to create autologous urethral constructs for the repair of urethral strictures.

DETAILED DESCRIPTION:
This is a Phase I clinical study to determine the safety and efficacy of using autologous, engineered urethral constructs for the treatment of urethral strictures in adult males.

The proposed study design is a prospective non-randomized and uncontrolled single-center investigation. Autologous urothelial cells (UCs) and smooth muscle cells (SMCs), obtained from enrolled male subjects' bladder tissue samples, will be culture expanded in vitro and used to seed tubular Polyglycolic Acid (PGA) scaffolds to create autologous urethral constructs for the repair of urethral strictures.

Male patients, aged 21-65 years old, seen in the Wake Forest Baptist Health urology clinic, referred to or self-referred to the study team, with recurrent urethral stricture, previously treated with dilation, internal urethrotomy, or urethroplasty, will be approached and offered consent to participate in in the trial. Up to 20 men may undergo screening procedures to identify 10 eligible subjects meeting all inclusion and exclusion criteria. All eligible subjects will undergo full thickness bladder tissue biopsies at Wake Forest Baptist Medical Center in Winston-Salem, North Carolina to obtain UCs and SMCs, which will be cultured and expanded and then seeded on tubular PGA scaffolds. Approximately 6 weeks after biopsy, the subjects will return to undergo surgical removal of the stricture and implant of the urethral construct. Subjects will be followed through 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Stricture of the urethra meeting the following criteria:

  a) History of at least one 15-60 mm in length, as determined by urethrography. c) Contains at least 1 strictured segment through which a 16 Fr flexible cystoscope cannot be atraumatically passed.
* Patients must be available for all follow-up visits.
* Ability to speak English.

Exclusion Criteria:

* Strictures of the meatus or prostatic urethra; any urethral stricture associated with or suspected to be urethral carcinoma, or strictures due to pelvic distraction injuries. Strictures <10 mm or >60 mm, as determined by urethrography, and criteria for bulbar urethral strictures excluding those with strictures <20 mm and >60 mm, as described by urethrography.
* Presence of untreated urinary tract infection.
* Presence or prior history of lichen sclerosis et atrophicus (previously termed 'balanitis xerotica obliterans').
* Uncontrolled bleeding disorder or patients with a platelet count less than 50,000, hemophilia or patients routinely receiving blood products for bleeding disorders.
* Any urological condition that would be likely to require additional urethral instrumentation during the period of investigation, including, but not limited to benign prostatic hyperplasia requiring treatment, use of alpha blockers, active prostate cancer, an unevaluated elevated prostate surface antigen (PSA), bladder cancer, or any recurrent urinary stone formation. Patients with evidence or diagnosis of any coagulation disorder (including concomitant anti-coagulation therapy at enrollment).
* Serum creatinine > 2.0 mg/dl or evidence of progressive renal disease.
* Patients with abnormal urologic conditions, including vesicoureteral reflux, bladder stones, bladder tumors and renal impairment.
* Subjects with an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >3 times the upper limit of normal.
* Subjects with an albumin value <3.0 g/dL.
* Subjects with uncontrolled diabetes, unstable cardiac and/or pulmonary disorders.
* Subjects with active tuberculosis (TB) requiring treatment in the past 3 years. Subjects with a current positive (≥5 mm induration for high-risk subjects; otherwise ≥10 mm of induration) purified protein derivative (PPD) test are excluded unless they have completed a full course of treatment for latent TB and have a negative chest x-ray film at enrollment.
* Subjects known to be colonized with either methicillin-resistant Staphylococcus aureus (MRSA) or vancomycin-resistant Enterococcus (VRE), or gentamicin-resistant organisms.
* Immunocompromised subjects or subjects receiving immunosuppressive agents (inhaled corticosteroids and chronic low-dose corticosteroids [≤0.25 mg/kg prednisone or equivalent per day] are permitted).
* Any history of alcohol and/or drug abuse.
* Current smoker.
* Documented history of, or positive result of HIV, Hepatitis B or C, or any infectious disease. External signs, sequelae, or positive serology of sexually transmitted disease (including HPV).
* Patients with a history of systemic conditions, including but not limited to HIV, diabetes and chronic liver disease (including Hepatitis B or C), that the Investigator believes may jeopardize the safety of the patient to participate in the study.
* Concurrent participation in any other clinical investigation during the period of this investigation. Patients who have been treated with any other investigational drug or participated in any investigational study within 30 days prior to enrollment in this study.
* Any current illness that might confound the results of this investigation, including but not limited to bladder atonia, neuropathic/neurogenic bladder, bladder outlet obstruction (other than urethral stricture), sphincteric dysfunction, or spinal cord injury.
* Any circumstance in which the investigator deems participation in the study is not in the subject's best interest.
* Inability to participate in all necessary study activities due to physical or mental limitations.
* Inability or unwillingness to return for all required follow-up visits.
* inability or unwillingness to sign informed consent.
* Patients requiring concomitant use of or treatment with immunosuppressive agents.
* Patients with neurological disorders (e.g., multiple sclerosis, Parkinson's disease).

Ages: 21 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of product-related, biopsy procedure-related, and injection procedure-related adverse events | monitored through 36 months post treatment
  Rate of adverse events reported for each patient

SECONDARY OUTCOMES:
Effectiveness of urethral construct in repairing urethral stricture | monitored through 36 months post construct implant
  Improvement in peak urinary flow rate defined as Qmax improvement from baseline

CONTACTS AND LOCATIONS:
Overall Officials: James Yoo, MD, Principal Investigator — Wake Forest Institute for Regenerative Medicine
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Wake Forest Institute for Regenerative Medicine (WFIRM), Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No